CLINICAL TRIAL: NCT02822118
Title: Therapeutic Effect of Chang'an I Recipe on Irritable Bowel Syndrome With Diarrhea: A Multicenter Randomized Double-Blind Placebo-Controlled Clinical Trial
Brief Title: Therapeutic Effect of Chang'an I Recipe on Irritable Bowel Syndrome With Diarrhea
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Xiyuan Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Digestion-03
Record Dates: First submitted 2016-06-27; First posted 2016-07-04 (Estimated); Last update posted 2016-09-05 (Estimated); Status verified 2016-06

CONDITIONS: Irritable Bowel Syndrome With Diarrhea
Keywords: IBS-D; Chang'an I Recipe; Placebo

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chang'an I Recipe (Experimental): Patients in this group were administered the Chang'an I Recipe for 8 weeks.
  Interventions: Drug: Chang'an I Recipe
- Placebo (Placebo Comparator): Patients in this group were administered the placebo for 8 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Chang'an I Recipe — Patients in this group were administered the Chang'an I Recipe, 150ml/bag, 3 times/day for 8 weeks.
  Other Names: The treatment group
  Arms: Chang'an I Recipe
Drug: Placebo — Patients in this group were administered the placebo, 150ml/bag, times/day for 8 weeks.
  Other Names: The control group
  Arms: Placebo

SUMMARY:
To evaluate the efficacy and safety of TCM decoction Chang'an I Recipe in the treatment of IBS-D. A multicenter, randomized, double-blind, placebo-controlled clinical trial was designed. Patients were applied for central random number and were given corresponding treatment according to inclusion sequences.The treatment group was administered the Chang'an I Recipe, 150ml/bag, 3 times/day; while the control group was administered the placebo, 150ml/bag, 3 times/day. Both courses of treatment were 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients meeting the diagnostic criteria of Western medicine for IBS-D;
* aged 18-70 years old; with a baseline IBS-SSS score over 75 points;
* voluntarily signed the informed consent;
* local resident who could ensure follow-ups, with basic reading ability.

Exclusion Criteria:

* Patients with IBS-C, -M, and uncertain forms;
* accompanied with serious lesions in major organs including heart, liver, and kidney, hematopoietic system diseases, and tumors;
* gastrointestinal organic disease (e.g., chronic pancreatitis), or systemic diseases affecting the digestive tract motion (e.g., hyperthyroidism, diabetes, chronic renal insufficiency, and nervous system diseases);
* undergoing or requiring constant use of drugs that may affect gastrointestinal functions (e.g., anti-cholinergic drugs, calcium channel blockers, 5-HT3 receptor antagonist, antidiarrheal agents, antacids, prokinetic agents, antidepressants, anxiolytics, and intestinal flora regulating drugs);
* with history of abdominal surgery (e.g., cholecystectomy);
* with an allergy history of tested drugs or severe allergy history of food;
* pregnant and lactating female;
* with a history of neurological or psychiatric disorders;
* or participating in other clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2013-01; Primary Completion 2015-12 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
change of Irritable Bowel Syndrome Symptom Severity Score (IBS-SSS) | IBS-SSS was evaluated by patients at 0, 2, 4 ,6 and 8 weeks.
  Score less than 75 points was considered as in remission, 75~175 as mild, 175~300 as moderate, and over 300 as severe.

SECONDARY OUTCOMES:
Serum markers regarding liver and kidney function | at baseline and 8 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: xudong Tang, Ph.D, Study Chair — XiYuan Hospital of China Academy of Traditional Chinese Medicine
Locations (5):
- China (5):
  - Xiyuan Hospital, Beijing, Beijing Municipality
  - Wangjing Hospital, Beijing, Beijing Municipality
  - Dongzhimen Hospital, Beijing, Beijing Municipality
  - Longhua Hospital, Shanghai, Shanghai Municipality
  - Zhejiang Provincial Hospital of TCM, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes